CLINICAL TRIAL: NCT03939312
Title: A Phase 3, Multicenter, Open-Label 40-week Extension Study to Evaluate the Long-Term Safety and Tolerability of Oral Atogepant for the Prevention of Migraine in Participants With Episodic Migraine
Brief Title: Extension Study to Evaluate the Long-Term Safety and Tolerability of Oral Atogepant for the Prevention of Migraine in Participants With Episodic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3101-309-002
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Episodic Migraine
Keywords: Migraine; Aura
MeSH Terms: conditions — Migraine Disorders; Epilepsy | interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atogepant 60 mg (Experimental): Participants received atogepant 60 mg, orally, once daily (QD) for up to 40 weeks.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Atogepant Tablets

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of atogepant 60 mg once a day for the prevention of migraine in participants with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and participant privacy information (eg, written authorization for use and release of health and research study information) obtained from the participant prior to initiation of any study-specific procedures.
* Participants must be using a medically acceptable and effective method of birth control during the course of the entire study.
* Eligible participants who completed the double-blind treatment period (Visit 7) and the follow-up period (Visit 8), if applicable, depending on the timing of study initiation, of Study 3101-301-002 (NCT03777059) without significant protocol deviations (eg, noncompliance to protocol-required procedures).

Exclusion Criteria:

* Female participant is pregnant, planning to become pregnant during the course of the study, or currently lactating. Women of childbearing potential must have a negative urine pregnancy test at Visit 1.
* Hypertension as defined by sitting systolic BP > 160 mm Hg or sitting diastolic BP > 100 mm Hg at Visit 1.
* Participants with clinically significant hematologic, endocrine, cardiovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Trugman, MD, Study Director — Allergan
Locations (112):
- United States (112):
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Alea Research, Phoenix, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Principals Research Group, Hot Springs, Arkansas
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Med Center Medical Clinic, Carmichael, California
  - Neuro Pain Medical Center, Fresno, California
  - California Headache and Balance Center, Fresno, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Paradigm Clinical Research Centers, Inc, La Mesa, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Long Beach Clinical Trials Services, Long Beach, California
  - Pharmacology Research Institute, Newport Beach, California
  - Newport Beach Clinical Research Associates, Newport Beach, California
  - Excell Research, Inc., Oceanside, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Desert Valley Research, Redlands, California
  - George J. Rederich, M.D. Inc., Redondo Beach, California
  - Optimus Medical Group, San Francisco, California
  - California Neuroscience Research, Sherman Oaks, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Aventura Neurological Associates, Aventura, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Sarkis Clinical Trials- Gainesville, Gainesville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Well Pharma Medical Research, Corp, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Sarasota Memorial Hospital Clinical Research Center, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Pediatric and Adolescent NeuroDevelopmental Associates (PANDA) Neurology, Atlanta, Georgia
  - Synexus Clinical Research, Inc, Atlanta, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Diamond Headache Clinic Ltd, Chicago, Illinois
  - JWM Neurology, Indianapolis, Indiana
  - Deaconess Clinic - Gateway Health Center, Newburgh, Indiana
  - PMG Research, Inc. d/b/a PMG Research of McFarland Clinic, Ames, Iowa
  - Heartland Research Associates, LLC, Newton, Kansas
  - College Park Family Care Center, Overland Park, Kansas
  - Collective Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, LLC - An AMR Company, Wichita, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - John R. Graham Headache Center Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Headache Center, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Synexus Clinical Research US, Inc., Omaha, Nebraska
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Piedmont Medical Research of Winston-Salem, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Ohio Clinical Research, LLC, Lyndhurst, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Jacob Murphy, Uniontown, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Partners in Clinical Research, LLC, Cumberland, Rhode Island
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Primary Care Associates/Synexus Clinical, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Hillcrest Family Practice, Simpsonville, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Psychiatry & Psychotherapy Partners Austin, Austin, Texas
  - Tekton Research, Austin, Texas
  - Synexus-US, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Centex Studies, Inc., Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Synexus Clinical Research, Inc, San Antonio, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Synexus-US, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc., South Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Sentara Neruology Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource and Core Clinical Research, Everett, Washington
  - Puget Sound Neurology, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Peterlin BL, Bond DS, Ailani J, Dodick DW, Liu Y, De Abreu Ferreira R, Smith JH, Dabruzzo B, Goadsby PJ, Trugman JM. Weight loss with atogepant during the preventive treatment of migraine: A pooled analysis. Cephalalgia. 2024 Dec;44(12):3331024241299753. doi: 10.1177/03331024241299753. PMID 39648629
- [Derived] Rizzoli P, Marmura MJ, Robblee J, McVige J, Sacco S, Nahas SJ, Ailani J, De Abreu Ferreira R, Ma J, Smith JH, Dabruzzo B, Ashina M. Safety and tolerability of atogepant for the preventive treatment of migraine: a post hoc analysis of pooled data from four clinical trials. J Headache Pain. 2024 Mar 11;25(1):35. doi: 10.1186/s10194-024-01736-z. PMID 38462625
- [Derived] Boinpally R, McNamee B, Yao L, Butler M, McGeeney D, Borbridge L, Periclou A. A Single Supratherapeutic Dose of Atogepant Does Not Affect Cardiac Repolarization in Healthy Adults: Results From a Randomized, Single-Dose, Phase 1 Crossover Trial. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1099-1107. doi: 10.1002/cpdd.940. Epub 2021 May 4. PMID 33942560
- [Derived] Min KC, Kraft WK, Bondiskey P, Colon-Gonzalez F, Liu W, Xu J, Panebianco D, Mixson L, Dockendorf MF, Matthews CZ, Boinpally R. Atogepant Is Not Associated With Clinically Meaningful Alanine Aminotransferase Elevations in Healthy Adults. Clin Transl Sci. 2021 Mar;14(2):599-605. doi: 10.1111/cts.12917. Epub 2020 Nov 24. PMID 33142014
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants rolled over from the lead-in study 3101-301-002 (NCT03777059) into this extension study. This study consisted of two periods: Open-label (OL) Treatment Period and Safety Follow-up Period.
Period: OL Treatment Period (40 Weeks)
Arm/Group | Atogepant 60 mg
Started | 685
Completed | 511
Not Completed | 174
Not completed — Withdrawal Criteria at Visit 1 | 43
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 35
Not completed — Lost to Follow-up | 19
Not completed — Pregnancy | 3
Not completed — Protocol Deviation | 16
Not completed — Non-compliance With Study Drug | 4
Not completed — Site Terminated by Sponsor | 3
Not completed — Reason Not Specified | 22
Period: Safety Follow-up 4 Weeks (Up to Week 44)
Arm/Group | Atogepant 60 mg
Started | 640 (Out of 685 participants, 640 participants who received treatment including 511 participants who completed the treatment entered safety follow-up period.)
Completed | 624
Not Completed | 16
Not completed — Withdrawal by Subject | 12
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of atogepant in this extension study.
Groups:
- Atogepant 60 mg: Participants received atogepant 60 mg, orally, QD for up to 40 weeks.
Arm/Group | Atogepant 60 mg
Number analyzed (Participants) | 685
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 604
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 631
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 86
  White | 578
  More than one race | 8
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Treatment-Emergent Adverse Event and Treatment-Emergent Serious Adverse Event (TEAEs/TESAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From dose of study drug until 30 days following last dose of study drug (up to approximately Week 44)
Population: Safety population included all participants who received at least 1 dose of atogepant in this extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg
Number analyzed (Participants) | 685
percentage of participants
  TEAEs | 62.5
  TESAEs | 3.4

2. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Laboratory Values as Assessed by the Investigator
Description: Clinical laboratory test values are considered PCS if they meet either the lower-limit or higher-limit PCS criteria defined in the categories below. Percentage of participants with PCS laboratory values are summarized for chemistry, hematology, and urinalysis. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during post-baseline are reported.
Time Frame: Up to Week 44
Population: Safety population included all participants who received at least 1 dose of atogepant in this extension study. Number analyzed are participants with data available for analyses of the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg
Number analyzed (Participants) | 685
percentage of participants
  Eosinophils Absolute Cell Count (10^9/L): > 2.0 × Upper Limit of Normal (ULN) | 0.3
  Hematocrit (Ratio): < 0.9 × Lower Limit of Normal (LLN): number analyzed (Participants) | 677
  Hematocrit (Ratio): < 0.9 × Lower Limit of Normal (LLN) | 1.5
  Hematocrit (Ratio): > 1.1 × ULN: number analyzed (Participants) | 677
  Hematocrit (Ratio): > 1.1 × ULN | 0.3
  Hemoglobin (g/L): < 0.9 × LLN: number analyzed (Participants) | 673
  Hemoglobin (g/L): < 0.9 × LLN | 2.2
  Lymphocytes Absolute Cell Count (10^9/L): < 0.7 × LLN: number analyzed (Participants) | 680
  Lymphocytes Absolute Cell Count (10^9/L): < 0.7 × LLN | 0.6
  Lymphocytes Absolute Cell Count (10^9/L): > 1.3 × ULN: number analyzed (Participants) | 680
  Lymphocytes Absolute Cell Count (10^9/L): > 1.3 × ULN | 0.3
  Monocytes Absolute Cell Count (10^9/L): < 0.5 × LLN: number analyzed (Participants) | 682
  Monocytes Absolute Cell Count (10^9/L): < 0.5 × LLN | 0.3
  Neutrophils Absolute Cell Count (10^9/L): < 0.7 × LLN: number analyzed (Participants) | 675
  Neutrophils Absolute Cell Count (10^9/L): < 0.7 × LLN | 1.6
  Neutrophils Absolute Cell Count (10^9/L): > 1.3 × ULN: number analyzed (Participants) | 675
  Neutrophils Absolute Cell Count (10^9/L): > 1.3 × ULN | 4.4
  Platelet Count (Thrombocytes) (10^9/L): < 0.5 × LLN: number analyzed (Participants) | 679
  Platelet Count (Thrombocytes) (10^9/L): < 0.5 × LLN | 0.1
  Platelet Count (Thrombocytes) (10^9/L): > 1.5 × ULN: number analyzed (Participants) | 679
  Platelet Count (Thrombocytes) (10^9/L): > 1.5 × ULN | 0.3
  Red Blood Cell Count (10^12/L): < 0.9 × LLN: number analyzed (Participants) | 679
  Red Blood Cell Count (10^12/L): < 0.9 × LLN | 2.4
  Red Blood Cell Count (10^12/L): > 1.1 × ULN: number analyzed (Participants) | 679
  Red Blood Cell Count (10^12/L): > 1.1 × ULN | 0.1
  White Blood Cell Count (10^9/L): < 0.9 × LLN: number analyzed (Participants) | 677
  White Blood Cell Count (10^9/L): < 0.9 × LLN | 3.5
  White Blood Cell Count (10^9/L): > 1.5 × ULN: number analyzed (Participants) | 677
  White Blood Cell Count (10^9/L): > 1.5 × ULN | 0.6
  Alanine Aminotransferase (SGPT) (U/L): ≥ 3.0 × ULN: number analyzed (Participants) | 682
  Alanine Aminotransferase (SGPT) (U/L): ≥ 3.0 × ULN | 0.3
  Aspartate Aminotransferase (SGOT) (U/L): ≥ 3.0 × ULN: number analyzed (Participants) | 683
  Aspartate Aminotransferase (SGOT) (U/L): ≥ 3.0 × ULN | 0.4
  Bicarbonate (HCO3) (mmol/L): < 0.9 × LLN: number analyzed (Participants) | 682
  Bicarbonate (HCO3) (mmol/L): < 0.9 × LLN | 0.7
  Bilirubin, Total (umol/L): ≥ 1.5 × ULN: number analyzed (Participants) | 682
  Bilirubin, Total (umol/L): ≥ 1.5 × ULN | 0.3
  Blood Urea Nitrogen (mmol/L): > 1.5 × ULN: number analyzed (Participants) | 682
  Blood Urea Nitrogen (mmol/L): > 1.5 × ULN | 0.1
  Creatine Kinase (U/L): > 2.0 × ULN: number analyzed (Participants) | 675
  Creatine Kinase (U/L): > 2.0 × ULN | 5.0
  Creatinine (umol/L): > 1.5 × ULN: number analyzed (Participants) | 683
  Creatinine (umol/L): > 1.5 × ULN | 0.4
  Glomerular Filtration Rate (GFR) Estimated Calculation (mL/min/1.73m^2): < 60 mL/min/1.73m^2: number analyzed (Participants) | 640
  Glomerular Filtration Rate (GFR) Estimated Calculation (mL/min/1.73m^2): < 60 mL/min/1.73m^2 | 15.6
  Glucose, Non-fasting (mmol/L): < 0.8 × LLN: number analyzed (Participants) | 672
  Glucose, Non-fasting (mmol/L): < 0.8 × LLN | 2.2
  Glucose, Non-fasting (mmol/L): > 2.0 × ULN: number analyzed (Participants) | 672
  Glucose, Non-fasting (mmol/L): > 2.0 × ULN | 0.9
  Phosphorus (mmol/L): < 0.9 × LLN: number analyzed (Participants) | 679
  Phosphorus (mmol/L): < 0.9 × LLN | 1.6
  Phosphorus (mmol/L): > 1.1 × ULN: number analyzed (Participants) | 679
  Phosphorus (mmol/L): > 1.1 × ULN | 0.6
  Potassium (mmol/L): > 1.1 × ULN: number analyzed (Participants) | 676
  Potassium (mmol/L): > 1.1 × ULN | 2.2
  Protein, Total (g/L): < 0.9 × LLN: number analyzed (Participants) | 682
  Protein, Total (g/L): < 0.9 × LLN | 0.7
  Uric Acid (Urate) (umol/L): > 1.2 × ULN: number analyzed (Participants) | 682
  Uric Acid (Urate) (umol/L): > 1.2 × ULN | 0.7
  Urine Glucose: At Least 1+: number analyzed (Participants) | 670
  Urine Glucose: At Least 1+ | 0.9
  Urine Protein: At Least 1+: number analyzed (Participants) | 648
  Urine Protein: At Least 1+ | 27.6

3. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Electrocardiograms (ECGs) Findings as Assessed by the Investigator
Description: 12-lead ECGs were performed at select study visits. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to Week 40
Population: Safety population included all participants who received at least 1 dose of atogepant in this extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg
Number analyzed (Participants) | 665
percentage of participants
  QRS Duration, Single Beat (msec): ≥ 150 milliseconds (msecs) | 0.3
  PR interval, Single Beat (msec): ≥ 250 msecs | 0.5
  QTcB interval, Single Beat (msec): > 500 msecs | 0.2
  QTcB interval, Single Beat (msec): Increase > 60 msecs | 0.3
  QTcF interval, Single Beat (msec): Increase > 60 msecs | 0.2
  QTcF interval, Single Beat (msec): >450 msecs | 3.4
  QTcF interval, Single Beat (msec): >480 msecs | 0.1

4. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Vital Sign Measurements as Assessed by the Investigator
Description: PCS postbaseline vital sign values are summarized for categories: systolic and diastolic blood pressures [sitting and standing], pulse rate [sitting and standing], respiratory rate, temperature, weight. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to Week 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg
Number analyzed (Participants) | 685
percentage of participants
  Systolic Blood Pressure Sitting (mmHg): ≤ 90 and Decrease of ≥ 20 | 1.9
  Systolic Blood Pressure Standing (mmHg): ≤ 90 and Decrease of ≥ 20 | 0.7
  Systolic Blood Pressure Standing (mmHg): ≥ 180 and Increase of ≥ 20 | 0.1
  Standing - Sitting Systolic Blood Pressure (mmHg): ≤ -20: number analyzed (Participants) | 673
  Standing - Sitting Systolic Blood Pressure (mmHg): ≤ -20 | 9.8
  Diastolic Blood Pressure Sitting (mmHg): ≤ 50 and Decrease of ≥ 15 | 0.6
  Diastolic Blood Pressure Sitting (mmHg): ≥ 105 and Increase of ≥ 15 | 1.0
  Diastolic Blood Pressure Standing (mmHg): ≤ 50 and Decrease of ≥ 15 | 0.7
  Diastolic Blood Pressure Standing (mmHg): ≥ 105 and Increase of ≥ 15 | 1.5
  Standing - Sitting Diastolic Blood Pressure (mmHg): ≤ -15: number analyzed (Participants) | 675
  Standing - Sitting Diastolic Blood Pressure (mmHg): ≤ -15 | 7.4
  Pulse Rate Sitting (beats/min): ≤ 50 and Decrease of ≥ 15 | 0.3
  Pulse Rate Standing (beats/min): ≤ 50 and Decrease of ≥ 15 | 0.4
  Pulse Rate Standing (beats/min): ≥ 120 and Increase of ≥ 15 | 1.8
  Standing - Sitting Pulse Rate (beats/min): ≥ 25: number analyzed (Participants) | 676
  Standing - Sitting Pulse Rate (beats/min): ≥ 25 | 6.8
  Weight (kg): Decrease of ≥ 7 percent (%) | 23.9
  Weight (kg): Increase of ≥ 7% | 9.2

5. Secondary Outcome: Number of Participants With Suicidal Ideation and Behaviour Using 5-Point Scale of Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. Suicidal ideation: Minimum total score 1, maximum total score 5; higher total scores indicate more suicidal ideation. Suicidal behavior: Minimum total score 0, maximum total score 4; higher total scores indicate more suicidal behavior.
Time Frame: OL Treatment Period: Up to Week 40; Safety Follow-up Period: Week 44
Population: Safety population included all participants who received at least 1 dose of atogepant in this extension study. One Safety population was used for the entire study. If participants were eligible for the Safety Follow-up they were included in the analyses even if they did not participate in the Safety Follow-up Period.
Measure: Count of Participants; unit: Participants
Groups:
- Atogepant 60 mg: Participants received atogepant 60 mg, orally, QD for up to 40 weeks in the open-label treatment period.
- Safety Follow-up Period: Following the open-label treatment period, participants entered the 4-week safety follow-up period.
Arm/Group | Atogepant 60 mg | Safety Follow-up Period
Number analyzed (Participants) | 685 | 685
Participants
  Suicidal Ideation | 4 | 1
  Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: From dose of study drug until 30 days following last dose of study drug (up to approximately Week 44)
Arm/Group | Atogepant 60 mg
All-Cause Mortality (participants affected / at risk) | 0/685
Serious Adverse Events (participants affected / at risk) | 23/685
Other Adverse Events (participants affected / at risk) | 71/685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atogepant 60 mg (N=685)
Gastritis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Concussion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple sclerosis (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Victim of abuse (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atogepant 60 mg (N=685)
Upper respiratory tract infection (Infections and infestations) | 38
Urinary tract infection (Infections and infestations) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03939312/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03939312/SAP_001.pdf